CLINICAL TRIAL: NCT01727856
Title: An Evaluation of a Novel Motion Tracking Enabled Knee Physical Therapy Application With Healthy Patients to Assess Reliability and Usability
Brief Title: Usability and Reliability of a New Physical Therapy Tool
Status: Completed | Type: Observational
Sponsor: Reflexion Health, Inc. (Industry)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: NMCSD.2012.0060; NIH CTSA 8KL2TR000110-05 (Other Grant/Funding Number: NIH CTSA 8KL2TR000110-05)
Record Dates: First submitted 2012-11-01; First posted 2012-11-16 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Normals
Keywords: rehabilitation; physical therapy; telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rehabilitation Measurement Tool: This single arm consists of all subjects which will interact with the tool under invstigation.
  Interventions: Device: Rehabilitation Measurement Tool

INTERVENTIONS:
Device: Rehabilitation Measurement Tool — The Rehabilitation Measurement Tool represents a telerehabilitation tool for physical therapy.

SUMMARY:
Rehabilitation exercise conducted at home following injury improves clinical and functional outcomes. Optimum compliance with prescribed exercise regimens requires regular patient instruction, performance assessment, monitoring and general encouragement from healthcare staff. Exercise at home though convenient for patients is not conducive for provision of the professional support needed to maximize prescribed regimen effectiveness.

Software in development by Reflexion Health Inc. along with the Naval Medical Center San Diego (NMCSD) is being designed to facilitate remote staff-patient interaction during at-home rehabilitative exercise sessions. Microsoft Kinect® will serve as the hardware platform for the designed software package tentatively called, "Reflexion." Kinect® contains a marker-less/controller-less motion tracking camera. The final Reflexion software will rely on a "Rehabilitation Measurement Tool (RMT)" to detect cardinal plane skeletal joint movement and its velocity utilizing the embedded Kinect® camera while also providing patient visual feedback via an avatar on a television screen.

In this observational minimal risk study, RMT/Kinect® functional reliability and usability will be assessed. Twenty healthy subjects will physically set-up and turn-on the hardware/software system; receive exercise directions from the RMT; then conduct a series of knee exercises similar to those prescribed after anterior cruciate ligament (ACL) repair.

An initial limited data set, obtained by Reflexion Health, provided validity and reliability measures. Eighteen degrees of absolute difference was detected between manual goniometry and Kinect® measurements in relevant planes of movement utilized during prescribed ACL exercise. Good relative agreement between RMT and goniometry scores was obtained (ICC = 0.89). A correctable systematic bias toward underestimation by the RMT will allow for future more accurate estimations of joint positioning improving face validity.

RMT functional reliability and general usability will be expressed in this study utilizing descriptive statistics and scaled questionnaires. Hardware component malfunction (Kinect® camera, laptop, PC, or LCD television/monitor) as well as RMT internally logged software errors and failure will tallied and measured to ascertain RMT reliability.

User-RMT interaction quality will be evaluated with video recordings of each set-up and exercise session. Specifically, usability measures will include: need for additional assistance setting-up or operating the RMT; number of attempts required by the subject to interact with a specific feature: time spent on specific elements during the session. Participant feedback will be elicited post-session using two scaled questionnaires: System Usability Scale (SUS)and Reflexion Usability Scale (RUS). Findings from the study will guide software modifications needed prior to implementation of future clinical studies within the NMCSD population.

DETAILED DESCRIPTION:
1. General Approach:

   We plan on using an observational study design to assess the reliability and usability of the RMT by healthy volunteers as they participate in a simulated session of knee physical therapy as presented by the RMT. Each session will be supervised by research staff and recorded for later review and assessment of areas of concern for reliability and usability.
2. Methods:

   The study will use 20 (n=20) healthy volunteers. These subjects will be actively recruited from Naval Medical Center San Diego and Orthopedic by research staff. We will also use an informational flyer placed in the NMCSD Physical Therapy and Orthopedic outpatient clinic waiting room. No medical records will be used to identify subjects for recruitment. Subjects will be approached by research staff and will be asked about participation and will undergo standard practices regarding meeting, inclusion and exclusion criteria and clinical trial consent by trained research staff. Those who consent to participate will be taken to an area that houses the RMT hardware and software. Subjects will then undergo a brief 5 minute tutorial on the setup, power-on, and navigation of the hardware and gesture controlled software.

   After the orientation session each subject will be presented the RMT hardware and asked to connect the hardware components via provided cables and subsequently power on the system and application as well as position themselves correctly in front of the camera. Next, they will be instructed to follow the on screen prompts to enter their subject ID and pertinent login information and navigate the system using gestures. Following the setup process they will then proceed to engage in four exercises sequentially presented by the RMT software. Approximately 5 repetitions of each exercise will be recorded and evaluated by the RMT after which the subject will be asked to follow the onscreen prompts to review a summary of their activity as presented by the RMT and exit the application. After their interaction with the RMT they will be asked to complete a System Usability Scale questionnaire as well as a Reflexion Usability Scale questionnaire.

   We anticipate the total time required by each subject will be approximately 45 minutes. Research staff will be available to provide any assistance as requested by the subjects in their interaction with the RMT. Additionally, staff will also intervene while consented subjects perform the exercises if they detect any signs of impending injury or harm. Subjects will be allowed to terminate their involvement at any time and for any reason.

   Review of the research staff notes during the subject interaction with the RMT, SUS and RUS results, and videotape of the interaction between the subject and RMT will be corroborated post-hoc.
   1. Sample Size

      We estimate the sample size of this study to be approximately 20 subjects. Since no direct comparison is being made to a control cohort, no inferential statistical analysis will be performed. This means that there is no meaningful way to appropriately power the study via sample size adjustments. Our choice of 20 subjects, therefore, was based on balancing the logistics required to test this platform with collecting sufficient data to understand the usability of then system.
   2. Randomization

      N/A
   3. Blinding

      N/A
   4. Initial Orientation Session

   Subjects will be given a brief video tutorial on how to connect the Kinect camera to the television and laptop, power on the RMT and Kinect camera, and operate the RMT hardware and software by research staff; any questions will be answered at that time regarding RMT operation. Then, subjects will be evaluated by a licensed, currently practicing physical therapist and shown the four exercises they will perform in the session. The therapist will work with each of the patients until they achieve a satisfactory performance in each of the exercises, as assessed by the therapist.
3. Components

   * Hardware:

     * Kinect Camera
     * LCD Television
     * Laptop PC
   * Software:

     * Windows 7 Operating System
     * Rehabilitation Measurement Tool Software Application
4. Statistical Analysis:

The primary goal of this research is to understand the usability and reliability of the system. Since the present application is relatively novel, there are no standard mthods to 'success' or 'failure' of the system. Therefore, we do not intend to perform any inferential statistical analyses. Rather, we will generate descriptive statistics to be used in a post-hoc fashion to determine system reliability, and usability for future applications to sick patients undergoing physical therapy for post-ACL reconstruction surgery. Descriptive statistics provide better insight into the data allowing a more informed assessment of potential risks of the system. Understanding the distributional nature of the data (e.g., normal symmetric, normal skewed, bimodal, etc.) and the variability of the data scores can better identify overall safety risks as well as help to specify individuals that could potentially incur a greater safety risk, should one exist.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Males and Females
* Age 18-35

Exclusion Criteria:

* Active knee symptoms
* Enrollment in knee physical therapy within 3 months of evaluation
* External or implanted lower extremity prosthetics
* Administration of regularly scheduled pain medication for lower extremities including oral, topical, or intra-articular routes of delivery
* Surgery or procedures within 3 months prior to enrollment
* Previous History of traumatic Knee Injury that required surgical intervention and/or resulted in baseline knee functional disability
* Pregnant women
* Significant cognitive impairment
* Neurovestibular deficits resulting in impaired balance and proprioception
* Traumatic brain injury
* Loss of function or immobilization of both upper extremities

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy males and femailes, ages 18-35
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Reliability | 30 minutes, patients followed for duration of set-up, initialization, and completion of RMT exercise protocol
  We have designed and plan to implement a measure, which quantifies the length of time for the subject to set-up and initialize the system which will be used to test inter-reliability of patients using the Reflexion Measurement Tool to complete the exercise protocol. After the patient completes the exercise protocol we will ask the patient to complete the Reflexion Usability Scale to provide their user feedback and experience.

SECONDARY OUTCOMES:
Usability | 30 minutes, patients followed for duration of set-up, initialization, and completion of RMT exercise protocol
  The number of interactions required by the study coordinator in order for the subject to correctly set up, initialize and complete the set protocol of physical therapy exercises using the Rehabilitation Measurement Tool. The study coordinator will use the Reflexion Usability Scale to quantify and measure outcome while subject is using the system to complete the exercise protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

REFERENCES:
- [Background] Hurley MV, Walsh NE, Mitchell H, Nicholas J, Patel A. Long-term outcomes and costs of an integrated rehabilitation program for chronic knee pain: a pragmatic, cluster randomized, controlled trial. Arthritis Care Res (Hoboken). 2012 Feb;64(2):238-47. doi: 10.1002/acr.20642. PMID 21954131
- [Background] Jan MH, Hung JY, Lin JC, Wang SF, Liu TK, Tang PF. Effects of a home program on strength, walking speed, and function after total hip replacement. Arch Phys Med Rehabil. 2004 Dec;85(12):1943-51. doi: 10.1016/j.apmr.2004.02.011. PMID 15605331
- [Background] Jette DU, Jette AM. Physical therapy and health outcomes in patients with knee impairments. Phys Ther. 1996 Nov;76(11):1178-87. doi: 10.1093/ptj/76.11.1178. PMID 8911431
- [Background] Harris GR, Susman JL. Managing musculoskeletal complaints with rehabilitation therapy: summary of the Philadelphia Panel evidence-based clinical practice guidelines on musculoskeletal rehabilitation interventions. J Fam Pract. 2002 Dec;51(12):1042-6. PMID 12540330
- [Background] Fischer DA, Tewes DP, Boyd JL, Smith JP, Quick DC. Home based rehabilitation for anterior cruciate ligament reconstruction. Clin Orthop Relat Res. 1998 Feb;(347):194-9. PMID 9520889
- [Background] Campbell R, Evans M, Tucker M, Quilty B, Dieppe P, Donovan JL. Why don't patients do their exercises? Understanding non-compliance with physiotherapy in patients with osteoarthritis of the knee. J Epidemiol Community Health. 2001 Feb;55(2):132-8. doi: 10.1136/jech.55.2.132. PMID 11154253
- [Background] Jette AM, Rooks D, Lachman M, Lin TH, Levenson C, Heislein D, Giorgetti MM, Harris BA. Home-based resistance training: predictors of participation and adherence. Gerontologist. 1998 Aug;38(4):412-21. doi: 10.1093/geront/38.4.412. PMID 9726128
- [Background] Fitzgerald GK. Therapeutic exercise for knee osteoarthritis: considering factors that may influence outcome. Eura Medicophys. 2005 Jun;41(2):163-71. PMID 16200033
- [Background] Pisters MF, Veenhof C, van Meeteren NL, Ostelo RW, de Bakker DH, Schellevis FG, Dekker J. Long-term effectiveness of exercise therapy in patients with osteoarthritis of the hip or knee: a systematic review. Arthritis Rheum. 2007 Oct 15;57(7):1245-53. doi: 10.1002/art.23009. PMID 17907210
- [Background] Rand D, Kizony R, Weiss PT. The Sony PlayStation II EyeToy: low-cost virtual reality for use in rehabilitation. J Neurol Phys Ther. 2008 Dec;32(4):155-63. doi: 10.1097/NPT.0b013e31818ee779. PMID 19265756
- [Background] Burke, J. W. et al. Optimising engagement for stroke rehabilitation using serious games. Vis Comput 25, 1085-1099 (2009).
- [Result] Pisters MF, Veenhof C, Schellevis FG, Twisk JW, Dekker J, De Bakker DH. Exercise adherence improving long-term patient outcome in patients with osteoarthritis of the hip and/or knee. Arthritis Care Res (Hoboken). 2010 Aug;62(8):1087-94. doi: 10.1002/acr.20182. PMID 20235201
- [Result] Zhiqiang Luo; Chee Kian Lim; Weiting Yang; Ke Yen Tee; Kang Li; Chao Gu; Kim Doang Nguen; I-Ming Chen; Song Huat Yeo; ,
- [Result] Zhou, H. Human motion tracking for rehabilitation--A survey. Biomedical Signal Processing and Control (2008).
- [Result] Papastergiou, M. Exploring the potential of computer and video games for health and physical education: A literature review. Computers & Education 53, 603-622 (2009).
- [Result] Broeren J, Claesson L, Goude D, Rydmark M, Sunnerhagen KS. Virtual rehabilitation in an activity centre for community-dwelling persons with stroke. The possibilities of 3-dimensional computer games. Cerebrovasc Dis. 2008;26(3):289-96. doi: 10.1159/000149576. Epub 2008 Jul 31. PMID 18667809
- [Result] Yu, C. A Study on Technology Acceptance of Applying Wii to Physical Therapy. (2008).
- [Result] Lange, B., Flynn, S. & Rizzo, A. Initial usability assessment of off-the-shelf video game consoles for clinical game-based motor rehabilitation. Phys. Ther. Rev. 14, 355-363 (2009).
- [Result] Clark R, Kraemer T. Clinical use of Nintendo Wii bowling simulation to decrease fall risk in an elderly resident of a nursing home: a case report. J Geriatr Phys Ther. 2009;32(4):174-80. doi: 10.1519/00139143-200932040-00006. PMID 20469567
- [Result] Holden, M., Dyar, T. & Schwamm, L. Home-based telerehabilitation using a virtual environment system. (2003)
- [Result] Rizzo AA, Strickland D, Bouchard S. The challenge of using virtual reality in telerehabilitation. Telemed J E Health. 2004 Summer;10(2):184-95. doi: 10.1089/tmj.2004.10.184. PMID 15319048
- [Result] Gövercin, M., Missala, I. M., Marschollek, M. & Steinhagen-Thiessen, E. Virtual Rehabilitation and Telerehabilitation for the Upper Limb. GeroPsych: The Journal of Gerontopsychology and Geriatric Psychiatry 23, 79-90 (2010).
- [Result] Sigal, L. Articulated Pose Estimation and Tracking: Introduction. Visual Analysis of Humans (2011).
- [Result] Lange, B., Rizzo, S., Chang, C. & Suma, E. Markerless Full Body Tracking: Depth-Sensing Technology within Virtual Environments. The Interservice/Industry , Simulation & Education Conference (I/ITSEC) (2011).
- [Result] Lewis GN, Woods C, Rosie JA, McPherson KM. Virtual reality games for rehabilitation of people with stroke: perspectives from the users. Disabil Rehabil Assist Technol. 2011;6(5):453-63. doi: 10.3109/17483107.2011.574310. Epub 2011 Apr 17. PMID 21495917
- [Result] Rand, D., Kizony, R., Feintuch, U. & Katz, N. Comparison of two VR platforms for rehabilitation: video capture versus HMD. … Teleoperators & Virtual Presence, Vol. 14, No. 2, April 2005, 147-160 (2005). 28. Mumford, N. et al. 2008 Virtual Rehabilitation. 2008 Virtual Rehabilitation 175-180 (2008).
- [Result] Kizony, R., Katz, N. & Tamar Weiss, P. L. Adapting an immersive virtual reality system for rehabilitation. J. Visual. Comput. Animat. 14, 261-268 (2003).
- [Result] Bruun, A. Evaluating the Usability of Home Healthcare Applications. Human-Centered Design of E-Health (2010).
- [Result] Gruchmrnann T. The impact of usability on patient safety. Biomed Instrum Technol. 2005 Nov-Dec;39(6):462-5. doi: 10.2345/0899-8205(2005)39[462:TIOUOP]2.0.CO;2. No abstract available. PMID 17432472
- [Result] Fairbanks RJ, Wears RL. Hazards with medical devices: the role of design. Ann Emerg Med. 2008 Nov;52(5):519-21. doi: 10.1016/j.annemergmed.2008.07.008. Epub 2008 Aug 22. No abstract available. PMID 18722693